CLINICAL TRIAL: NCT02434601
Title: Dentin Treatments for Restorations of Cervical Lesions Non-carious: a Randomized Clinical Trial of Three Years
Brief Title: Dentin Treatments for Restorations of Cervical Lesions Non-Carious
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Rafael Guerra Lund, Professor, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Federal University of Pelotas
Record Dates: First submitted 2015-03-04; First posted 2015-05-05 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-04

CONDITIONS: Adhesion
Keywords: Non-carious cervical lesions; Randomized clinical trial; Permanent dental restoration; Dentin; Adhesion; Restoration; Sensitivity; Prophylaxis; Randomized
MeSH Terms: conditions — Tissue Adhesions; Hypersensitivity | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment of Dentin Surface (Other): Treatment of Dentin Surface: Restoration made following the protocol recommended by the manufacturer of the materials.
  Interventions: Procedure: Treatment of Dentin Surface
- Dentin Surface (Experimental): Treatment of Dentin Surface: Increased etching dentin for 15 seconds to 30 seconds
  Interventions: Procedure: Dentin Surface
- Treatment (Experimental): Treatment of Dentin Surface: Intervention with the cavity prophylaxis probe ultrasound blunt applied for 30 seconds in Surface hypermineralized non-carious dentin cervical lesions. Therefore, the restoration was done following the protocol recommended by the manufacturer of the material.
  Interventions: Procedure: Treatment

INTERVENTIONS:
Procedure: Treatment of Dentin Surface — * Experimental Group 1: Increase the etching time to 30 seconds, performed with phosphoric acid gel at 37%, prior to application of the resin adhesive.
  * Experimental Group 2: Prophylaxis cavity probe / blunt tip of ultrasound, applied for 30 seconds on the dentin surface hypermineralized of cervical lesions non-carious.
  Both restorative procedures were performed using a conventional adhesive system and composite restorative nanoparticulate.
  Other Names: Preconditioning of Dental Surface
  Arms: Treatment of Dentin Surface
Procedure: Dentin Surface — Treatment of Dentin Surface: Increased etching dentin for 15 seconds to 30 seconds
  Arms: Dentin Surface
Procedure: Treatment — Treatment of Dentin Surface: Intervention with the cavity prophylaxis probe ultrasound blunt applied for 30 seconds in Surface hypermineralized non-carious dentin cervical lesions. Therefore, the restoration was done following the protocol recommended by the manufacturer of the material.
  Arms: Treatment

SUMMARY:
The surface of non-carious cervical lesions (LCNC) is a challenge to adhesive systems, it presents a dentin layer sclera hypermineralized, presence of bacteria and lack of mechanical retention, so this study aimed to evaluate the influence of different surface treatments on LCNC through a randomized clinical trial. Patients with LCNC were referred to the study and selected according to the inclusion criteria, such as the presence of at least 3 LCNC. Three different types of surface treatment were carried out in LCNC: control group, 15 seconds of etching dentin; Group I, acid etching of dentin in 30 seconds; and group II, cavity prophylaxis with ultrasound for 30 seconds. The remaining steps of the adhesive and restorative procedure was the same for all groups, following the material manufacturer's recommendations. Evaluations of restorations will be carried out in periods of one week (baseline), six months, one year, two years and three years as of tooth sensitivity, integrity and color change. Data will be analyzed by McNemar and chi-square test.

DETAILED DESCRIPTION:
Ethical considerations This study was designed and conducted according to the guidelines Consolidated Standards of Reporting of Trials (CONSORT) for the preparation of randomized controlled clinical trials (Altman et al., 2001), after approval by the Research Ethics Committee (protocol number CEP-035 -2011- FO / UFPel), Faculty of Dentistry, Federal University of Pelotas - RS / Brazil.

Study design

Calculation for determining the sample

Based on the literature, the sample size was obtained assuming an average annual rate of failure 6% for Class V restorations performed with conventional adhesive systems (PEUMANS et al., 2005b), with 80% power and significance level of 5%. From the recommendations of the American Dental Association (2010), we estimated an annual failure rate of 12% for restorations in relative isolation. For this, a sample of 28 was determined by monitoring patients for a minimum of 5 years, considering possible attrition of 20%.

Recruitment and selection of patients The search strategy of individuals interested in participating in this clinical trial was conducted through the dissemination of the project through the display of posters and distribution of pamphlets in FO / UFPEL as well as in basic health units (BHU) located in the urban area Pelotas. In addition, the study had the collaboration of students representatives of class associations, coordinating teachers of clinical activities and dentists the public health system, to increase the receptivity and the accession of potential volunteers.

All patients were referred, or directly sought dental care, with diagnosis of non-carious cervical lesion, were scheduled for evaluation exam.

Two students of the seventh semester, under the supervision of the responsible of this study, carried out the consultations on the premises of FO / UFPEL. Initially, the presence of LCNC was assessed by visual inspection with wooden spatula aid. If so, we filled out a patient's medical record, containing identification data, general and dental history. In addition, the dental chart was performed using mirror, explorer, millimeter periodontal probe, clinical tweezers, cotton rolls and saliva sucker. From the clinical examination, the LCNC were sorted review of its features. The dentin sensitivity was evaluated by applying air jet for 3 seconds, the distance 2-3 cm of the labial surface, and sensitivity degree record from a visual analogue scale. Likewise, the pulpal vitality was visualized using cotton balls previously moistened with the gas jet cooling at -50 ° C.

Patients who met the inclusion and exclusion criteria received an information letter about the nature and proposal of the study. After reading, we asked the volunteers to sign a consent form and informed about their participation.

In a second clinic session, the patients underwent a process of adaptation of oral health for the prevention, control, removal of plaque and dental calculus. Professional intervention consisted in scraping, smoothing and polishing dental, using curettes / periodontal files, glass / rubber cone, Robinson brush, prophylaxis paste and contra angle low speed.

Operator training Six candidates for operators (students between the seventh and eighth semester of FOUFPEL) participated in a training process to ensure the standardization of clinical procedures and minimize the variation of different operators.

First stage (theoretical): A lecture was given, lasting about two hours, consisting in the presentation of materials and techniques for the removal or modification of hypermineralized surface layer of dentin-carious cervical lesions. It was also performed routine detailed statement to be instituted during the sessions. A manual containing the material operating instructions and the protocol of clinical procedures, was made available to students.

Second stage (practice): Students went through pre-clinical activities, watching the demonstration and subsequently performing Class V restorations on mannequins. Secondly, they performed the same procedures for volunteers who, despite presenting LCNC with restorative needs, were not included in this study. Therefore, such patients received restorative treatment under conditions identical to the patients involved in the study, but not part of the sample.

At the end of training and calibration steps, the functions of the working group delegated by using the performance of individual students as selection criteria. Were chosen two operators, who have restorative procedures, and two assistants to support operators and completion of medical records. The other students were in charge of sterilization of instruments, scheduling appointments, molding, photographic record, oral hygiene orientation, periodontal treatment, among other dental procedures offered to patients. All the above mentioned steps were performed under direct supervision of the responsible for the study.

Preparation of the patient: Four weeks before the start of the study, the patients were subjected to a sweep session, smoothing and polishing supragingival. In addition, patients received individualized instruction for mechanical control of dental biofilm, including guidance on the brushing technique and flossing. During the monitoring period, was also offered dental support to patients involved in the study.

Clinical Protocol Initially, prophylaxis element to be restored was made with glass and rubber based slurry of pumice and water. Then the color of the restoration was selected with the aid of a color scale (Vitapan Classical, Vita Zahnfabrik, Bad Säckingen, Germany). Local anesthesia was Also, when necessary. In the same query, the patient received restorative action in three LCNC to submit clinical features compatible. Randomization as the technique for the surface layer removal or modification hypermineralized to be applied in each place by drawing lots. The restorations were initiated by the previous LCNC, with the priority needs, the main complaint: aesthetic, functional aspects and / or symptoms such as tooth sensitivity, etc. Each patient had to have at least 3 teeth to be restored because of the 3 types of treatments employed. It draw lots 3 treatments individually for each tooth. For example, if a patient possessed the three lesions selected, the drawing is performed to be selected for each tooth treatment be subjected to a treatment. If the patient possess more than 3 lesions was performed again for the draw element 4 and so on with the other.

We emphasize also that each operator held the same number of restorative interventions, and one was prepared following the protocol recommended by the manufacturer of the materials, another increasing the etching time to 30 seconds on dentin and finally the third cavity was restored after performing a cavity prophylaxis with ultrasound probe applied for 30 seconds. The remaining steps were carried out following the protocol recommended by the manufacturer of restorative materials employed.

The rubber dam was accomplished through the use of lip retractor, wire retractor # 000 (Ultrapak Cord, Ultradent, South Jordam, UT, USA), cotton rolls and saliva sucker. The first element to be introduced in the oral cavity was the lip retractor, printing expulsion lips and cheeks. Cotton rolls were positioned in the upper labial sulcus at the lower labial sulcus and in the sublingual region, to absorb the saliva flow coming mainly from the major salivary glands. The retractor wire is inserted into the gingival sulcus with the aid of blunt spatula, without generating excessive pressure in the periodontium.

Prior to the implementation of restoration, there has been no type of cavity preparation, or beveling of cavosurface margins. However, each LCNC dentin surface was subjected to various removal or modification of the techniques hypermineralized ultra-surface layer, as follows:

* Control Group: Restoration made following the protocol recommended by the manufacturer of the materials;
* Experimental Group 1: Increase the etching time to 30 seconds, performed with phosphoric acid gel at 37%, prior to application of the resin adhesive. The following steps to acid etching followed the protocol recommended by the manufacturer of the materials;
* Experimental Group 2: Prophylaxis cavity with ultrasound probe, applied for 30 seconds on the dentin surface hypermineralized of cervical lesions non-carious. Soon after, the restoration was made following the protocol recommended by the manufacturer of the materials.

Both restorative procedures were performed using a conventional adhesive system (Single Bond II, 3M ESPE, St. Paul, MN, USA) and composite restorative nanoparticulate (Filtek Z350, 3M ESPE, St. Paul, MN, USA), closely following the operating instructions provided by the manufacturer. The restorations were placed by incremental technique using about 2 or 3 increments restorative composite, as the size of LCNC. The increments were taken and adapted to the cavity starting with the margin in enamel with spatulas, brushes and siliconadas tips for composite resin. An LED device with minimum intensity 1450 mW / cm2 was used for polymerization.

Finally, the finish of the restoration was performed by using # 12 scalpel blade, diamond and fine-grained multi-laminated drills, in order to remove excess material and / or improve the shape of the contour restorations. The polishing of the same was done with employment siliconadas tips, floppies sandpaper (Sof-Lex Pop-On, 3M ESPE, St. Paul, MN, USA), felt-specific folders and polishing discs.

Reviews of restorations Two examiners (graduated in Dentistry) will go through a training process and calibration until present intra agreement index and inter-examiner of at least 80%. In the event of disagreement as to the assessment criteria, the same terião to get a consensus through direct revaluation of restorations and / or by means of digital photographs.

After the training phase and calibration, the evaluators 'blind', ie without any involvement with the conditions which patients will be submitted, shall proceed independently, clinical evaluations of restorations. At this time, the evaluators will use magnifying glass, mirror, explorer, millimeter periodontal probe, clinical tweezers, cotton rolls and saliva sucker. Data relating to dentin sensitivity and pulp vitality will also be collected through the air jet application and application cotton balls have been wetted with gas jet cooling to -50 ° C, respectively. Digital photographs will also be consulted by the evaluators.

The properties will be evaluated sensitivity, color change and integrity of the restoration.

Statistical analysis Clinical evaluations will occur in the following periods: 1 week (baseline), six months, a year, two years and three years after insertion of the restorations using the evaluated criteria. The data will be tabulated and submitted to statistical analysis, considering 80% power and 5% significance level.

Will be held descriptive analysis with calculation of ratios to characterize the sample and dental restorations. To compare outcomes in the pre- and post-intervention according to the treatment groups and also the comparison of outcome between treatment groups will be used chi-square test and McNemar test. The analyzes will be performed using Stata 12.1 software.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least three non-carious cervical lesions on the buccal aspect of previous vital teeth or premolars;
* Visible plaque index presence and / or gingival bleeding index of at most 20%;
* Probing depth of at least 3 mm in the experimental site and / or buccal 4 mm in any place;
* Patients with good general health condition;
* Patients able to understand and sign the letter of information and the free and informed consent;
* Patients willing to return every six months to revaluation queries.

Exclusion Criteria:

* Presence of less than 20 teeth in the mouth;
* Patients undergoing orthodontic treatment;
* Patients with occlusion problems;
* Veneers with wear over 50% of the incisal / occlusal structure;
* Absence of tooth antagonist.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-03 (Actual); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Number of teeth with lost restorations | From Baseline restorations at 3 years

SECONDARY OUTCOMES:
Presence or not of marginal leakage | From Baseline restorations at 3 years
Presence or not of dentin hypersensitivity | From Baseline restorations at 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Rafael G Lund, PhD, Principal Investigator — Federal University of Pelotas

REFERENCES:
- [Result] Demarco FF, Baldissera RA, Madruga FC, Simoes RC, Lund RG, Correa MB, Cenci MS. Anterior composite restorations in clinical practice: findings from a survey with general dental practitioners. J Appl Oral Sci. 2013 Nov-Dec;21(6):497-504. doi: 10.1590/1679-775720130013. PMID 24473714
- [Result] Akimoto N, Takamizu M, Momoi Y. 10-year clinical evaluation of a self-etching adhesive system. Oper Dent. 2007 Jan-Feb;32(1):3-10. doi: 10.2341/06-46. PMID 17288322
- [Result] Bartlett D, Ganss C, Lussi A. Basic Erosive Wear Examination (BEWE): a new scoring system for scientific and clinical needs. Clin Oral Investig. 2008 Mar;12 Suppl 1(Suppl 1):S65-8. doi: 10.1007/s00784-007-0181-5. Epub 2008 Jan 29. PMID 18228057
- [Result] Bartlett DW, Lussi A, West NX, Bouchard P, Sanz M, Bourgeois D. Prevalence of tooth wear on buccal and lingual surfaces and possible risk factors in young European adults. J Dent. 2013 Nov;41(11):1007-13. doi: 10.1016/j.jdent.2013.08.018. Epub 2013 Sep 1. PMID 24004965
- [Result] Hickel R, Roulet JF, Bayne S, Heintze SD, Mjor IA, Peters M, Rousson V, Randall R, Schmalz G, Tyas M, Vanherle G. Recommendations for conducting controlled clinical studies of dental restorative materials. Clin Oral Investig. 2007 Mar;11(1):5-33. doi: 10.1007/s00784-006-0095-7. Epub 2007 Jan 30. PMID 17262225
- [Result] Karakaya S, Unlu N, Say EC, Ozer F, Soyman M, Tagami J. Bond strengths of three different dentin adhesive systems to sclerotic dentin. Dent Mater J. 2008 May;27(3):471-9. doi: 10.4012/dmj.27.471. PMID 18717178
- [Result] Kim SY, Lee KW, Seong SR, Lee MA, Lee IB, Son HH, Kim HY, Oh MH, Cho BH. Two-year clinical effectiveness of adhesives and retention form on resin composite restorations of non-carious cervical lesions. Oper Dent. 2009 Sep-Oct;34(5):507-15. doi: 10.2341/08-006C. PMID 19830963
- [Result] Lopes GC, Baratieri CM, Baratieri LN, Monteiro S Jr, Cardoso Vieira LC. Bonding to cervical sclerotic dentin: effect of acid etching time. J Adhes Dent. 2004 Spring;6(1):19-23. PMID 15119583
- [Result] Lopes GC, Vieira LC, Monteiro S Jr, Caldeira de Andrada MA, Baratieri CM. Dentin bonding: effect of degree of mineralization and acid etching time. Oper Dent. 2003 Jul-Aug;28(4):429-39. PMID 12877429
- [Result] Moretto SG, Russo EM, Carvalho RC, De Munck J, Van Landuyt K, Peumans M, Van Meerbeek B, Cardoso MV. 3-year clinical effectiveness of one-step adhesives in non-carious cervical lesions. J Dent. 2013 Aug;41(8):675-82. doi: 10.1016/j.jdent.2013.05.016. Epub 2013 Jun 6. PMID 23747824
- [Result] Perdigao J. Dentin bonding-variables related to the clinical situation and the substrate treatment. Dent Mater. 2010 Feb;26(2):e24-37. doi: 10.1016/j.dental.2009.11.149. Epub 2009 Dec 14. PMID 20005565
- [Result] Peumans M, Kanumilli P, De Munck J, Van Landuyt K, Lambrechts P, Van Meerbeek B. Clinical effectiveness of contemporary adhesives: a systematic review of current clinical trials. Dent Mater. 2005 Sep;21(9):864-81. doi: 10.1016/j.dental.2005.02.003. PMID 16009415
- [Result] Ritter AV, Heymann HO, Swift EJ Jr, Sturdevant JR, Wilder AD Jr. Clinical evaluation of an all-in-one adhesive in non-carious cervical lesions with different degrees of dentin sclerosis. Oper Dent. 2008 Jul-Aug;33(4):370-8. doi: 10.2341/07-128. PMID 18666493
- [Result] Da Rosa Rodolpho PA, Donassollo TA, Cenci MS, Loguercio AD, Moraes RR, Bronkhorst EM, Opdam NJ, Demarco FF. 22-Year clinical evaluation of the performance of two posterior composites with different filler characteristics. Dent Mater. 2011 Oct;27(10):955-63. doi: 10.1016/j.dental.2011.06.001. Epub 2011 Jul 16. PMID 21762980
- [Result] Salz U, Bock T. Testing adhesion of direct restoratives to dental hard tissue - a review. J Adhes Dent. 2010 Oct;12(5):343-71. doi: 10.3290/j.jad.a19741. PMID 20978636
- [Result] Tay FR, Pashley DH. Resin bonding to cervical sclerotic dentin: a review. J Dent. 2004 Mar;32(3):173-96. doi: 10.1016/j.jdent.2003.10.009. PMID 15001284
- [Result] Wilder AD Jr, Swift EJ Jr, Heymann HO, Ritter AV, Sturdevant JR, Bayne SC. A 12-year clinical evaluation of a three-step dentin adhesive in noncarious cervical lesions. J Am Dent Assoc. 2009 May;140(5):526-35. doi: 10.14219/jada.archive.2009.0220. PMID 19411519